CLINICAL TRIAL: NCT02619747
Title: A Multi-centre, Randomised, Open Label, Placebo-controlled, Two-period Crossover Study to Evaluate 4-hour Esophageal pH Change in GERD Patients After Administration of Compound Sodium Alginate Oral Suspension Sachets or Placebo Sachets
Brief Title: Compound Sodium Alginate Oral Suspension Sachet 4-hour Esophageal pH Study in GERD Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Problems with recruitment
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GA1218
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Gastro-esophageal Reflux Disease (GERD)
Keywords: pH monitoring
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compound Sodium Alginate Oral Suspension sachet (Active Comparator): Single dose of contents of two 10 ml sachets of Compound Sodium Alginate Oral Suspension
  Interventions: Drug: Compound Sodium Alginate Oral Suspension sachet; Drug: Matched placebo
- Matched placebo (Placebo Comparator): Single dose of contents of two 10 ml sachets of matched placebo
  Interventions: Drug: Compound Sodium Alginate Oral Suspension sachet; Drug: Matched placebo

INTERVENTIONS:
Drug: Compound Sodium Alginate Oral Suspension sachet
  Other Names: Gaviscon sachets
Drug: Matched placebo

SUMMARY:
Multi-centre, randomised, open-label, placebo-controlled, two-period crossover study of 4 hour pH monitoring following a refluxogenic meal and drink.

DETAILED DESCRIPTION:
This is a multi-centre, randomised, open-label, placebo-controlled, two-period crossover study. After signing a written informed consent (ICF), patients will undergo a screening period of up to 10 days (Visit 1) which will require the patient to return to the clinic on several occasions. At the start of the screening process patients will have 24 hour (h) pH monitoring which will include one standardised refluxogenic meal after a 4 h fast. The 24 h pH monitoring results will be used as a key criteria for patient eligibility and to provide the patients with diagnostic information on their symptoms. After 24 h pH monitoring, eligible patients will be supplied with Compound Sodium Alginate Oral Suspension sachet to take as required for symptom relief between visits (up to 2×10ml sachets four times daily: 30 minutes after breakfast, 30 minutes after lunch, 30 minutes after dinner and immediately before lying down for bed, stopping dosing at least 24 hours prior to Visit 2).

Patients who satisfy the study entry requirements within 10 days of consent, will be randomised to receive either two Compound Sodium Alginate Oral Suspension sachets (2×10ml) or two placebo sachets (2×10ml) following placement of a pH electrode after a 4 h fast and a standardised refluxogenic meal at Visit 2.

Upon completion of the Visit 2 4-hour post-dose pH monitoring period patients will be re-supplied with Compound Sodium Alginate Oral Suspension sachets to take as required for symptom relief (up to 2×10ml sachets four times daily: 30 minutes after breakfast, 30 minutes after lunch, 30 minutes after dinner and immediately before lying down for bed, stopping dosing at least 24 hours prior to Visit 3) for 7 ± 2 days. Patients will return for Visit 3 after 7 ± 2 days. Visit 3 will consist of repeat pH catheter insertion (4 hour fast followed by refluxogenic test meal consumption) and pH monitoring, receiving the alternative randomised treatment at Visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis: Current evidence of symptomatic GERD in accord with the Montreal definition. Patients should have a GERD history of frequent episodes of GERD-related symptoms during at least the last 2 months prior to study screening. The patient must also meet the following criteria:

  * The main symptom is heartburn and/or acid reflux. Symptoms persist or have occurred repeatedly for at least the last 2 months;
  * The frequency of occurrence of heartburn is ≥ 3 days/week and the score of severity of heartburn in general is moderate or severe within 3 weeks before screening
* Patients who are willing to consume the entire standard refluxogenic test meal.
* Patients who have a screening 24 h pH monitoring test assessing the percentage of time when the pH falls below pH 4 which confirms significant acid reflux of >4.2% over the 24 h period.

Exclusion Criteria:

* Patients who have a history of drug, solvent or alcohol abuse (weekly alcohol intake ≥ 140g).
* Patients who have suffered cardiac chest pain within the last year.
* Patients who have suffered a recent, significant unexplained weight loss of more than 6 kg in the last 6 months.
* Female patients of childbearing potential who, for the duration of the study, are either unwilling or unable to take adequate contraceptive precautions or are unwilling to be sexually abstinent.
* Pregnancy or lactating mother.
* Patients with a history and/or symptom profile suggestive of the following: any other gastrointestinal (GI) disease (e.g. gastric or duodenal erosions and polyps larger than 0.5 cm), erosive GERD Los Angeles [LA] classification grades C-D, Barrett's esophagus, acute peptic ulcer and/or ulcer complications, Zollinger-Ellison syndrome, gastric carcinoma, pyloric stenosis, oesophageal or gastric surgery, intestinal obstruction, current pernicious anaemia, hiatal hernias greater than 3 cm, requirement for low sodium diet, known gastrointestinal bleeding (hematochezia or hematemesis) within the last 3 months, and severe diseases of other major body systems.
* Patients who have taken anti-cholinesterase drugs, traditional Chinese medicines for treating gastrointestinal disease, sucralfate or misoprostol preparations within 7 days prior to screening or throughout the study.
* Patients who have taken Proton Pump Inhibitors (PPIs) during the 28 days prior to screening, prokinetics or H2 antagonists during the 5 days prior to screening, or systemic glucocorticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs except low dose aspirin given for cardioprotection) on more than 3 consecutive days during the last 28 days prior to screening.
* Patients who have taken any antacids within 24 hours before screening (Visit 1) and throughout the remainder of the study.
* Patients taking mucous membrane protection drugs or motility stimulants for 5 days prior to screening and throughout the study.
* Patients who are vegetarian.
* Patients with difficulty in swallowing.
* Patients with known hypophosphataemia, phenylketonuria or hypercalcaemia.
* Patients who have previously undergone esophageal, gastric or duodenal surgery at any time or who have undergone any other major surgery with general anaesthesia within the last three months.
* Patients with severe constipation, or history of intestinal obstruction.
* In the opinion of the Investigator, patients with insufficient heart or kidney function and patients who require a low sodium diet.
* Patients either with any co-existing condition which, in the opinion of the Investigator, would be likely to compromise patient safety or interfere with assessment of efficacy; or with any clinically significant abnormal laboratory values.
* Patients with impaired renal function or severe renal insufficiency.
* Any previous history of allergy or known intolerance to any of the formulation constituents
* Clinically significant abnormalities in the physical examination, electrocardiogram (ECG) and safety analysis.
* Patients taking or requiring to take macrolide antibiotics, such as erythromycin, azithromycin, from the day before screening.
* Previously randomised into the study.
* Employee at study site.
* Partner or first-degree relative of the Investigator.
* Participation in a clinical study in the previous 6 months.
* Unable in the opinion of the Investigator to comply fully with the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of time during the 4 hour post dosing period with pH below pH 4. | 4 hours post-dose

SECONDARY OUTCOMES:
Percentage of time during the 4 hour post dosing period with pH below pH 5 | 4 hours post-dose
Number of occasions during the 4 hour post dosing period when pH falls below pH 4 | 4 hours post-dose
Number of occasions during the 4 hour post dosing period when pH falls below pH 5 | 4 hours post-dose
Number of reflux episodes during the 4 hour post dosing period with pH below pH 4 for at least 5 minutes | 4 hours post-dose
Percentage of time during the first hour post dosing with pH below pH 4 | 1 hour post-dose
Percentage of time during the first hour post dosing with pH below pH 5 | 1 hour post-dose
Number of occasions during the first hour post dosing when pH falls below pH 4 | 1 hour post-dose
Number of occasions during the first hour post dosing when pH falls below pH 5 | 1 hour post-dose
The longest reflux time during the 4 hour post dosing period | 4 hours post-dose
DeMeester score | 4 hours post-dose
Overall proportion of patients with adverse events (AEs) | 20 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affilated Hospital Sun Yat-Sen University, Guangzhou, Guangdong, China